CLINICAL TRIAL: NCT02630563
Title: A Study of the Safety, Tolerability and Pharmacokinetics of Oral CellCept® (Mycophenolate Mofetil, MMF) in Pediatric Liver Transplant Recipients on Concomitant Treatment With Cyclosporine and Corticosteroids
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral CellCept (Mycophenolate Mofetil) in Pediatric Liver Transplant Recipients on Concomitant Treatment With Cyclosporine and Corticosteroids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to extremely slow recruitment, infrequent use of combination triple therapy (MMF, cyclosporine, steroids), study was discontinued; Part 2 was not conducted.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA16497
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric Liver Transplantation
MeSH Terms: interventions — Adrenal Cortex Hormones; Cyclosporine; Mycophenolic Acid

ARMS (1):
- Mycophenolate Mofetil+Corticosteroids+Cyclosporine (Experimental): Part 1: Participants will receive mycophenolate mofetil. Part 2: Participants will receive mycophenolate mofetil along with cyclosporine and corticosteroids.
  Interventions: Drug: Corticosteroids; Drug: Cyclosporine; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: Corticosteroids — Corticosteroids will be administered as per center practice. The choice of corticosteroid drug will also be based on center practice.
Drug: Cyclosporine — Cyclosporine will be administered as per center practice.
Drug: mycophenolate mofetil — Part 1: Mycophenolate mofetil will be administered as per center practice. Part 2: Mycophenolate mofetil will be administered as per dose determined in Part 1.
  Other Names: CellCept

SUMMARY:
The study is planned to be conducted in 2 parts. The first part (open label, multi-center, non-controlled) of the study will estimate a dose that would provide a mycophenolic acid (MPA) exposure in pediatric participant that is comparable to that achieved in adult liver transplant participants receiving the approved dose of mycophenolate mofetil (MMF, CellCept). The second part (open-label, multi-center, single-arm Phase IV study) of the study will provide the pharmacokinetics, efficacy and safety profile of the proposed dose in the immediate post-transplant period. This study will be conducted at two centers based in the United States of America. Twelve pediatric transplant participants receiving a first liver allograft from a cadaveric or living donor will be enrolled in this study. Stable pediatric liver transplant participants who are at least 6 months post-transplant and who were already receiving stable dose of MMF in combination with cyclosporine will be enrolled into the study. Participants should have received stable MMF dose according to center practice for at least seven days in order to get steady state pharmacokinetics (PK). Participants also should have received stable concomitant doses of cyclosporine (for at least 2 days) and corticosteroids per center practice. Participants will be aged between 9 months and 12 years, with at least 6 participants greater than or equal to (>/=) 9 months and less than (<) 36 months, of whom at least 2 will be <24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be between 3 months and 12 years of age
* Participant is a recipient of a first liver allograft from cadaveric or living donors
* Participant is a single-organ recipient (liver only)
* Female participants of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli International Units per milliliter (mIU/mL) within one week prior to PK sampling
* Female participants of childbearing potential must use two reliable forms of contraception simultaneously unless abstinence is the chosen method
* Effective contraception must be used before beginning of PK sampling
* Participants must be able to receive oral medication
* Participants must be at least 6 months post-transplant and had started on MMF in the early post-transplant period (within 2 weeks of transplant)
* Participants must be receiving stable doses of MMF per center practice for at least 7 days prior to PK sampling
* In addition, participants must be receiving stable doses of cyclosporine and corticosteroids, according to center practice
* Participants' parent/guardian are capable of understanding the purposes and risks of the study and must sign an informed consent for the study

Exclusion Criteria:

* Pregnant or nursing adolescents
* Participants who had undergone dialysis within two weeks before PK sampling
* Participants with active systemic infections
* Participants with absolute neutrophil counts (ANC) of less than 1300 per microliter (µL), or platelets counts less than 50 000/µL or hemoglobin at a concentration below a set lower limit (according to center practice, but not less than 8 grams per deciliter) at the time of study entry
* Participants with active peptic ulcer disease
* Participants with severe diarrhea (more than 5 watery stools per day) or other gastrointestinal disorders which might interfere with their ability to absorb oral medication
* History of positive human immunodeficiency virus (HIV) test

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2003-05; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (2):
- United States (2):
  - San Francisco, California
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 02 May 2003 and 20 January 2005. This study was conducted at 2 sites in United States (US). Overall, 9 participants entered the study.
Pre-assignment Details: Thirty five participants were screened; 9 entered the study following a screening period of up to 14 days. Stable pediatric liver transplant participants who were at least 6 months post-transplant and who were receiving stable dose of Mycophenolate Mofetil (MMF) in combination with cyclosporine were enrolled into the study.
Groups:
- Drug MMF: Participants receiving drug MMF twice daily along with stable concomitant doses of cyclosporine (for at least 2 full days) and corticosteroids as per center practice for at least 7 days prior to Pharmacokinetic (PK) sampling were observed up to Day 16
Period: Overall Study
Arm/Group | Drug MMF
Started | 9
Completed | 8
Not Completed | 1
Not completed — Administrative | 1

BASELINE CHARACTERISTICS:
Population: All Patient Population included all participants who were enrolled in the trial
Arm/Group | Drug MMF
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4

OUTCOME MEASURES:

1. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0-12 Hours for Mycophenolic Acid and Mycophenolic Acid Glucuronide Phenolic Glucuronide of Mycophenolic Acid
Description: The area under the plasma concentration-time curve from time zero to twelve hours (AUC [0-12h]) is area under the plasma concentration-time curve from time zero through 12 hours. AUC (0-12) hours was computed using the linear trapezoidal rule. For the calculations of AUC (0-12h), concentrations below the limit of quantification were assigned a value of zero if they occurred at the beginning of a profile. When such values appeared at the end of a profile they were assigned as missing data. AUC was reported in microgram hour per milliliter (mcg*h/mL).
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 4.0, 8.0, and 12.0 hours post oral dosing for participants greater than (>) 24 months, and at pre-dose, 0.75, 2.0, 4.0 and 12.0 hours post oral dosing for participants less than (<) 24 months
Population: The PK population included all randomized and replaced participants adherent to the PK section of the protocol
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Drug MMF
Number analyzed (Participants) | 8
mcg*h/mL
  MPA Raw | 29 (20.3)
  MPAG Raw | 487 (185)
  MPAG (MPA Equivalents) | 289 (109)

2. Secondary Outcome: Maximum Plasma Concentration for Mycophenolic Acid and Mycophenolic Acid Glucuronide
Description: The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration. Cmax was obtained directly from the measured plasma concentration-time curves.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 4.0, 8.0, and 12.0 hours post oral dosing for participants > 24 months, and at pre-dose, 0.75, 2.0, 4.0 and 12.0 hours post oral dosing for participants < 24 months
Population: The PK population was used for the analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Drug MMF
Number analyzed (Participants) | 8
mcg/mL
  MPA Raw | 7.98 (3.69)
  MPAG Raw | 54.6 (26.8)
  MPAG (MPA Equivalents) | 32.4 (15.9)

3. Secondary Outcome: Time to Maximum Plasma Concentration for Mycophenolic Acid and Mycophenolic Acid Glucuronide
Description: Tmax is the amount of time after dosing to when the maximum concentration of MPA and MPAG was achieved.
Time Frame: as for outcome 2
Population: The PK population was used for the analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Drug MMF
Number analyzed (Participants) | 8
hour
  MPA Raw | 1.35 [0.5 to 2.03]
  MPAG Raw | 1.99 [1.52 to 4.13]

4. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event.
Time Frame: Up to Day 32
Population: The safety population included all participants who were enrolled in the trial
Measure: Number; unit: participants
Arm/Group | Drug MMF
Number analyzed (Participants) | 9
participants
  Participants with AE | 1
  Participants with SAE | 0

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 12 Hours of Mycophenolic Acid Normalized for Dose And for Body Surface Area
Description: The area under the plasma concentration-time curve from time zero to twelve hours (AUC [0-12h]) is area under the plasma concentration-time curve from time zero through 12 hours. AUC (0-12) hours was computed using the linear trapezoidal rule. For the calculations of AUC (0-12h), concentrations below the limit of quantification were assigned a value of zero if they occurred at the beginning of a profile. When such values appeared at the end of a profile they were assigned as missing data. AUC0-12h was normalized to 600 milligram per square meter (mg/m^2) and 1.5 gram. AUC was reported in microgram hour per milliliter (mcg*h/mL).
Time Frame: as for outcome 1
Population: The pharmacokinetic (PK) population included all randomized and replaced participants adherent to the PK section of the protocol.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Drug MMF
Number analyzed (Participants) | 8
mcg*h/mL
  Normalized to 600mg/m^2 | 65.6 (56.2)
  Normalized to 1.5g | 363 (360)

6. Secondary Outcome: Plasma Concentration of Mycophenolic Acid and Its Metabolite Mycophenolic Acid Glucuronide at Each Time Point
Description: Mycophenolic Acid Glucuronide (MPAG) is an active metabolite of Mycophenolic Acid (MPA).
Time Frame: as for outcome 1
Population: The PK population included all randomized and replaced participants adherent to the PK section of the protocol.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Drug MMF
Number analyzed (Participants) | 8
mcg/mL
  Raw MPA at 0.0 | 0.786 (0.681)
  Raw MPA at 0.50 | 9.03 (4.34)
  Raw MPA at 0.75 | 5.67 (3.14)
  Raw MPA at 1.00 | 5.84 (3.13)
  Raw MPA at 1.50 | 6.16 (5.08)
  Raw MPA at 2.00 | 6.23 (4.54)
  Raw MPA at 4.00 | 1.89 (1.90)
  Raw MPA at 8.00 | 1.38 (1.72)
  Raw MPA at 12.00 | 0.676 (0.795)
  Raw MPAG at 0.00 | 26.2 (20.4)
  Raw MPAG at 0.50 | 26.5 (1.13)
  Raw MPAG at 0.75 | 45.8 (28.2)
  Raw MPAG at 1.00 | 37.2 (4.81)
  Raw MPAG at 1.50 | 43.2 (12.9)
  Raw MPAG at 2.00 | 51.0 (27.9)
  Raw MPAG at 4.00 | 46.3 (21.3)
  Raw MPAG at 8.00 | 19.2 (13.4)
  Raw MPAG at 12.00 | 14.6 (7.35)

ADVERSE EVENTS:
Time Frame: Up to Day 32
Description: All participants enrolled were included in the safety analysis.
Arm/Group | Drug MMF
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug MMF (N=9)
Pyrexia (General disorders) | 1

LIMITATIONS AND CAVEATS:
Part I of the study was terminated early with 9 participants enrolled (8 of which were evaluable for PK), and Part II of the study was not performed due to extremely slow recruitment and the infrequent use of the combination of triple therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.